CLINICAL TRIAL: NCT06643351
Title: Intrapartum Maternal Glucose Control and Effect on Neonatal Hypoglycemia
Brief Title: Intrapartum Glucose Control and Risk of Neonatal Hypoglycemia
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pittsburgh (Other)
Responsible Party: Principal Investigator, Praveen Ramesh, Fellow Physician, Division of Maternal-Fetal Medicine, Department of Obstetrics, Gynecology, and Reproductive Sciences, University of Pittsburgh
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: STUDY24050197
Record Dates: First submitted 2024-10-12; First posted 2024-10-16 (Actual); Last update posted 2025-12-15 (Actual); Status verified 2025-12

CONDITIONS: Gestational Diabetes Mellitus in Pregnancy; Pregestational Diabetes Mellitus; Neonatal Hypoglycemia
Keywords: Gestational Diabetes; Pregestational Diabetes; Neonatal Hypoglycemia; Intrapartum Glucose
MeSH Terms: conditions — Diabetes, Gestational

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Standard Intrapartum Glucose Target Range (Active Comparator): The goal intrapartum glucose target range will be 70-110mg/dl. Insulin infusion will be initiated when maternal capillary glucose exceeds 110 mg/dL.
  Interventions: Other: Standard Intrapartum Glucose Target Range
- Liberalized Intrapartum Glucose Target Range (Experimental): The goal intrapartum glucose target range will be 70-160mg/dl. Insulin infusion will be initiated when maternal capillary glucose exceeds 160 mg/dL.
  Interventions: Other: Liberalized Intrapartum Glucose Target Range

INTERVENTIONS:
Other: Standard Intrapartum Glucose Target Range — Intrapartum maternal glucose management involves frequent blood sugar checks and the use of insulin intravenous drip as needed. Maternal capillary blood sugar is checked every 4 hours in early labor, 2 hours in active labor and hourly during the second stage of labor. The frequency of maternal glucose monitoring will not differ by study group. The goal intrapartum glucose target range will be 70-110mg/dl. Insulin infusion will be initiated when maternal capillary glucose exceeds 110 mg/dL. Once an insulin infusion is initiated, glucose monitoring frequency will occur by protocol. A hypoglycemia protocol is initiated if the maternal blood sugar is less than 60mg/dl.
  Arms: Standard Intrapartum Glucose Target Range
Other: Liberalized Intrapartum Glucose Target Range — Intrapartum maternal glucose management involves frequent blood sugar checks and the use of insulin intravenous drip as needed. Maternal capillary blood sugar is checked every 4 hours in early labor, 2 hours in active labor and hourly during the second stage of labor. The frequency of maternal glucose monitoring will not differ by study group. The goal intrapartum glucose target range will be 70-160mg/dl. Insulin infusion will be initiated when maternal capillary glucose exceeds 160 mg/dL. Once an insulin infusion is initiated, glucose monitoring frequency will occur by protocol. A hypoglycemia protocol is initiated if the maternal blood sugar is less than 60mg/dl.
  Arms: Liberalized Intrapartum Glucose Target Range

SUMMARY:
The purpose of this study is to assess whether a liberal intrapartum glycemic target range compared to usual care standard control ranges will lead to a decrease in the rate of neonatal hypoglycemia among pregnant patients in labor with diabetes.

DETAILED DESCRIPTION:
Neonatal hypoglycemia is a leading cause of admission to the neonatal ICU (NICU) and is associated with increased costs, separation from mothers, and when severe, long term neurological sequelae. Prior research has suggested an association between intrapartum maternal glucose and the risk of neonatal hypoglycemia, so current insulin administration protocols aimed to maintain the blood glucose close to 100mg/dl.

However, recent studies have found inconsistent evidence of a relationship between intrapartum maternal glucose and neonatal hypoglycemia, Furthermore, on review of previously established protocols, improved maternal glucose control came with an increased frequency of neonatal hypoglycemia. Thus, these findings have suggested that relaxing the intrapartum goals for maternal glucose may be associated with improved neonatal outcomes.

Few randomized controlled trials (RCTs) exist in evaluating neonatal outcomes comparing liberal versus tight intrapartum glycemic control. Recent RCTs have found that tight maternal glucose control in labor was associated with lower mean neonatal blood glucose levels in the first 24 hours of life. While another recent RCT found that a permissive blood glucose (up to 180mg/dl) threshold was associated with equivalent neonatal blood glucose levels when compared to the standard, strict thresholds (up to 110mg/dl).

In this study, participants will be recruited at delivery planning outpatient visits or at admission to labor and delivery and stratified by type of diabetes into two groups, either Type 1 Diabetes or Gestational Diabetes(GDM)/Type 2 diabetes. They will then be randomized to one of two intervention groups. The liberalized treatment group will have a target Glucose Range 70 - 160mg/dl and receive treatment via insulin drip will be initiated if the blood sugar exceeds the upper bound. The standard treatment Group will have a glucose target Glucose Range 70 - 110mg/dl and receive treatment via insulin drip will be initiated if the blood sugar exceeds the upper bound.

The specific aim of this project is to determine the effectiveness of liberalized intrapartum glycemic targets in reducing the incidence of neonatal hypoglycemia.

ELIGIBILITY:
Inclusion Criteria:

* Pregnant patients with Pre-gestational (Type 1 or Type 2) or Gestational Diabetes
* Singleton Gestations
* Greater than or equal to 35 weeks gestation
* Planned for vaginal delivery at the University of Pittsburgh Medical Center Magee-Womens Hospital (UPMC MWH)

Exclusion Criteria:

* Major fetal anomalies anticipated to require NICU admission
* Planned Cesarean delivery

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 218 (Estimated)
Dates: Start 2024-12-03 (Actual); Primary Completion 2026-05 (Estimated); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
Immediate postnatal Neonatal hypoglycemia | Within the first 24 hours after delivery.
  Number of newborns with neonatal hypoglycemia, defined as a blood glucose of less than 45mg/dL

SECONDARY OUTCOMES:
Any neonatal hypoglycemia | Prior to neonatal discharge, up to 42 days after delivery.
  Number of newborns with neonatal hypoglycemia, defined as a blood glucose of less than 45mg/dL
Mean neonatal blood glucose | Prior to neonatal discharge, up to 42 days after delivery.
  Measured in mg/dL
Neonatal Hypoglycemia Requiring IV Treatment | Prior to neonatal discharge, up to 42 days after delivery.
  number of newborns with hypoglycemia that requires IV treatment
NICU admission | Prior to discharge, up to 42 days after delivery.
  Number of NICU admission for any indication.
Maternal Intrapartum Hyperglycemia | During labor( for up to 200 hours)
  Number of participants that have hyperglycemia episodes. Hyperglycemia is defined as blood sugar levels greater than 180 mg/dl
Maternal intrapartum hypoglycemia | During labor( for up to 200 hours)
  Number of participants that have hypoglycemia episodes. Hyp0glycemia is defined as blood sugar levels less than 60 mg/dl
Mean maternal intrapartum blood glucose | During labor( for up to 200 hours)
  Overall mean maternal glucose values in mg/dl

CONTACTS AND LOCATIONS:
Overall Officials: Praveen Ramesh, M.D., Principal Investigator — University of Pittsburgh
Locations (1):
- Magee-Women's Hospital of UPMC, Pittsburgh, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No
There is currently no plan to make individual participant data available to other researchers. The findings are anticipated to be reported in standard specialty journals.

REFERENCES:
- [Background] Dude AM, Niznik C, Peaceman AM, Yee LM. Evaluation of an Intrapartum Insulin Regimen for Women With Diabetes. Obstet Gynecol. 2020 Aug;136(2):411-416. doi: 10.1097/AOG.0000000000003940. PMID 32649492
- [Background] Yamamoto JM, Benham J, Mohammad K, Donovan LE, Wood S. Intrapartum glycaemic control and neonatal hypoglycaemia in pregnancies complicated by diabetes: a systematic review. Diabet Med. 2018 Feb;35(2):173-183. doi: 10.1111/dme.13546. PMID 29117445
- [Background] American College of Obstetricians and Gynecologists' Committee on Practice Bulletins-Obstetrics. ACOG Practice Bulletin No. 201: Pregestational Diabetes Mellitus. Obstet Gynecol. 2018 Dec;132(6):e228-e248. doi: 10.1097/AOG.0000000000002960. PMID 30461693
- [Background] Dude A, Niznik CM, Szmuilowicz ED, Peaceman AM, Yee LM. Management of Diabetes in the Intrapartum and Postpartum Patient. Am J Perinatol. 2018 Sep;35(11):1119-1126. doi: 10.1055/s-0038-1629903. Epub 2018 Mar 13. PMID 29534258
- [Background] Burns CM, Rutherford MA, Boardman JP, Cowan FM. Patterns of cerebral injury and neurodevelopmental outcomes after symptomatic neonatal hypoglycemia. Pediatrics. 2008 Jul;122(1):65-74. doi: 10.1542/peds.2007-2822. PMID 18595988